CLINICAL TRIAL: NCT03174704
Title: Longitudinal Determinants of Medication Adherence in COPD
Brief Title: Medication Adherence Research in COPD Patients
Acronym: MARC
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00091482; 1R01HL128620-01A1 (NIH)
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: COPD; Medication Adherence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is the third leading cause of death, affects over 24 million people in the US and is the leading cause of disability with projected healthcare costs at almost $50 billion. The goal of this study is to identify novel and potentially powerful targets for behavioral interventions in COPD which has been understudied despite its tremendous detrimental impact on overall public health.

DETAILED DESCRIPTION:
The Centers for Medicare and Medicaid Services (CMS) has specifically targeted COPD hospital readmissions as a meaningful quality outcome that could result in financial penalties highlighting the significant impact of COPD on our overall health system. The growing availability of efficacious medication, stands in stark contrast to the poor health outcomes experienced by COPD patients. One possible explanation for this gap is low rates of medication adherence; some studies report that only 25% of COPD patients take at least 80% of their prescribed medications. Pharmacy refill records indicate that adherence to COPD medications is significantly lower than adherence rates seen in other chronic illnesses including hypertension, diabetes, and congestive heart failure. Significant negative long term health outcomes may be magnified by non-adherence to prescribed medications in COPD.

This study proposes to systematically identify modifiable determinants of adherence in COPD based on the Theory of Self-Regulation in 360 patients with COPD. A novel and significant innovation of this study is the use of mobile health (mhealth) technology to objectively assess medication use. No previous study of self-regulation theory has utilized objective measure of adherence. A further innovation of the study is the use of ecological momentary assessment (EMA) of patient reported symptoms and beliefs to evaluate longitudinal associations between observation (patient symptoms) judgements (medication use to relieve symptoms), and reactions (self-efficacy, outcome expectancy, and medication beliefs) in real time. This study will be the first to objectively evaluate the application of the Self-Regulation Theory in COPD and to examine the long-term longitudinal impact of medication adherence on disease progression in a diverse sample.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* Physician diagnosis of COPD
* Prescribed a long-term controller medication for COPD
* Moderate COPD on the basis of meeting one of the following criteria:

  1. Gold Stage II-IV disease with forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) ≤70% and FEV1 (% predicted) <80% or
  2. One or more hospital admissions, two or more emergency department (ED) visits, or prescription of oral steroids for COPD exacerbation in the past 12 months or ever having used home oxygen
* Cognitive ability to provide informed consent

Exclusion Criteria:

- Non-English speaking

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll 360 patients (40 years of age or older) with physician diagnosed COPD and are prescribed a long-term controller medication for COPD
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | 5 years
  Measured by electronic medication monitoring

SECONDARY OUTCOMES:
% Predicted Forced Expiratory Volume (FEV) | 5 years
  Measured by spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Michelle N Eakin, Ph.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Christiana Care Health System, Newark, Delaware
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
We do not share individual participant data.